CLINICAL TRIAL: NCT06884722
Title: Social Perception and Dopaminergic Modulation in Patients With Parkinson's Disease: a Functional MRI Study (Park Social-E-Motion)
Brief Title: Brain Mechanisms of Social Perception in Parkinson's Disease
Acronym: Park Social
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 69HCL24_0681
Record Dates: First submitted 2025-03-07; First posted 2025-03-19 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Social Perception in Parkinson's Disease
Keywords: Functional MRI; Parkinson's disease; Social Cognition; Point light display
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: For patients: one MRI scan in the OFF dopaminergic treatment condition and one MRI scan in the ON dopaminergic treatment condition (randomized order by block).
  For controls: one MRI scan.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Stage 1: PD patients (Other): 20 adult patients with Parkinson disease will perform a behavioral task of social perception.
  Interventions: Behavioral: Behavioral task of social perception (stage 1); Other: Neurological and neuropsychological assessments; Other: Neurological assessments of Parkinson's disease symptoms and caregiver burden
- Stage 1: healthy volunteers (Other): 20 adult patients without neurologic disorders will perform a behavioral task of social perception.
  Interventions: Behavioral: Behavioral task of social perception (stage 1); Other: Neurological and neuropsychological assessments
- Stage 2: PD patients (Other): 23 adult patients with Parkinson disease will perform a behavioral task of social perception during functional MRI recording.
  Interventions: Other: Functional magnetic resonance imaging: 3 Tesla magnetic resonance imaging (stage 2); Other: Neurological and neuropsychological assessments; Other: Neurological assessments of Parkinson's disease symptoms and caregiver burden
- Stage 2: healthy volunteers (Other): 20 adult volunteers without neurologic disorder will perform a behavioral task of social perception during functional MRI recording
  Interventions: Other: Functional magnetic resonance imaging: 3 Tesla magnetic resonance imaging (stage 2); Other: Neurological and neuropsychological assessments

INTERVENTIONS:
Behavioral: Behavioral task of social perception (stage 1) — Patients with Parkinson disease and healthy volunteer are engaged in a social perception behavioral task.
  Arms: Stage 1: PD patients; Stage 1: healthy volunteers
Other: Functional magnetic resonance imaging: 3 Tesla magnetic resonance imaging (stage 2) — Patients with Parkinson disease and healthy volunteer are assessed by functional magnetic resonance imaging while they are engaged in a social perception behavioral task.
  2 times for patients with Parkinson disease (during ON-levodopa and OFF-levodopa) Once for healthy volunteer
  Arms: Stage 2: PD patients; Stage 2: healthy volunteers
Other: Neurological and neuropsychological assessments — Patients with Parkinson disease and healthy volunteer will undergo a neurological and neuropsychological assessment with several evaluations: weight, height, medical history, global cognitive performance (MoCA and BREF score), apathy (LARS score), depression (BDI-II score), social cognition (mini-SEA), and quality of life (PDQ39 self-questionnaire).
Other: Neurological assessments of Parkinson's disease symptoms and caregiver burden — Patients with Parkinson disease will undergo a neurological assessment of motor and non-motor symptoms of Parkinson's disease (MDS-UPDRS III & IV scale and MDS-NMS scale) and caregiver burden (Zarit scale).
  Arms: Stage 1: PD patients; Stage 2: PD patients

SUMMARY:
Social cognition is a complex process that enables humans to interpret social information and behave appropriately in a social environment. Social cognition can be impaired in Parkinson's disease patients, worsening quality of life and relationships with those around them, even at an early stage. These alterations are manifested in particular by impairments of the recognition of facial emotions and body movements, involving the motor system. The aim of this study is to understand the brain mechanisms associated with impaired social perception in people with Parkinson's disease using functional MRI and a behavioural task for the perception of social interaction scenes depicted by "Point Light Display" (PLD).This study will investigate the effect of dopaminergic modulation on the networks associated with the perception of movement and mirror system, the observation of action (parietal cortex, superior temporal sulcus), and those associated with the mentalization of others' cognitive or emotional states (prefrontal cortex and limbic system).

The study is thus divided into 2 stages.

* Stage 1 "preliminary": Preliminary validation of the experimental task
* Stage 2 "imagery": Assessment of brain activity (BOLD signal) related to social perception in imaging

ELIGIBILITY:
Inclusion Criteria:

* Male or female between 30 and 75 years of age
* Freely-given informed consent to participate to this study (written form)
* Affiliated with a social security system or equivalent;
* Person diagnosed with Parkinson's disease according to MDS-UPDRS criteria for at least 3 years and receiving dopaminergic treatment (e.g. : LEVODOPA, CARBIDOPA, BENZERASIDE, ENTACAPONE, MODOPAR, SINEMET, STALEVO, PRAMIPEXOLE, SIFROL, ROPINIROLE, REQUIP ; ROTIGOTINE, NEUPRO, PIRIBEDIL, TRIVASTAL, RASAGILINE, AZILECT, CONTAM, AMANTADINE, MANTADIX, APOMORPHINE, APOKINON, DOPACEPTIN, FOSLEVODOPA, FOSCARBIDOPA, SCYOVA) (for patients only)
* Effective contraception for women of childbearing age or post-menopausal women (only for patients and healthy volunteers in stage 2 "imaging")
* Requiring dopa testing as part of routine care (only for patients in stage 2 "imaging")
* No disabling cognitive impairment (MOCA score ≥ 26)
* No diagnosis of chronic disease associated with disability (only for healthy volunteers)

Exclusion Criteria:

* Contraindication to MRI (only for patients and healthy volunteers in step 2 "imaging"):

  * Wearing a pacemaker not approved for 3 Tesla MRI
  * Presence of intracerebral ferromagnetic or magnetizable material
  * Presence of intraocular ferromagnetic or magnetizable foreign bodies
  * Presence of non-removable ferro-magnetic or magnetizable foreign bodies in the cephalic region
  * Claustrophobia
* History of head trauma with loss of consciousness lasting more than 30 min (only for patients and healthy volunteers in step 2 "imaging")
* Participant not agreeing to be informed in the event of incidental discovery of an abnormality on MRI (only for patients and healthy volunteers in stage 2 "imaging")
* Tremor or disabling dyskinesias preventing MRI (only for patients in stage 2)
* Having exceeded the annual amount of compensation allowed for participation in research protocols (only for healthy volunteers)
* Pregnant, parturient or breast-feeding women
* Persons deprived of liberty by judicial or administrative decision
* Persons under psychiatric care
* Persons admitted to a health or social institution for purposes other than research
* Adults under legal protection (guardianship, curatorship)
* Participants in other intervention research involving a period of exclusion still in progress at the time of pre-inclusion.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 83 (Estimated)
Dates: Start 2025-07-15 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
BOLD signal difference in the brain networks associated with social perception in Parkinson's patients compared with age- and sex-matched healthy volunteers | Up to 75 days
  BOLD signal difference in the brain networks associated with social perception in Parkinson's patients compared with age- and sex-matched healthy volunteers during a social perception behavioural task using point light display

SECONDARY OUTCOMES:
BOLD signal difference in the brain networks associated with social perception in Parkinson's patients compared with age- and sex-matched healthy volunteers for the emotional valence | Up to 75 days
  BOLD signal difference in the brain networks associated with social perception in Parkinson's patients compared with age- and sex-matched healthy volunteers during a social perception behavioural task using point light display with emotional content
BOLD signal difference in the brain networks associated with social perception in Parkinson's patients in the OFF versus ON dopaminergic treatment conditions | Up to 75 days
  BOLD signal difference in the brain networks associated with social perception in Parkinson's patients during a social perception behavioural task using point light display in the OFF versus ON dopaminergic treatment conditions
BOLD signal difference in the brain networks associated with social perception in Parkinson's patients in the emotional content and OFF versus ON dopaminergic treatment conditions | Up to 75 days
  BOLD signal difference in the brain networks associated with social perception in Parkinson's patients during a social perception behavioural task using point light display for the emotional content and the OFF versus ON dopaminergic treatment conditions
Group correlation between clinical and neuropsychological scores and BOLD signal difference in patients with Parkinson's disease | Up to 75 days
  Group correlation between clinical and neuropsychological scores and BOLD signal difference in the brain networks associated with social perception in Parkinson's patients during a social perception behavioural task using point light display for the emotional content and the OFF versus ON dopaminergic treatment conditions
Group correlation between the integrity of substantia nigra and locus coeruleus nuclei measured on anatomical MRI and the BOLD signal difference in the brain networks associated with social perception in Parkinson's patients | Up to 75 days
  Group correlation between the integrity of substantia nigra and locus coeruleus nuclei measured on anatomical MRI and the BOLD signal difference in the brain networks associated with social perception in Parkinson's patients during a social perception behavioural task using point light display

CONTACTS AND LOCATIONS:
Locations (1):
- Service de neurologie - troubles du mouvement et pathologies neuromusculaires, Hôpital neurologique Pierre Wertheimer/GHE, Bron, France